CLINICAL TRIAL: NCT02688517
Title: Targeted Genomic Analysis of Human Cancers
Brief Title: Targeted Genomic Analysis of Blood and Tissue Samples From Patients With Cancer
Status: Recruiting | Type: Observational
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Rutgers Cancer Institute of New Jersey (Other)
Responsible Party: Principal Investigator, Shridar Ganesan, MD, PhD, Associate Professor of Medicine and Pharmacology Medical Oncology, Rutgers Cancer Institute of New Jersey
Other Study IDs: Pro2012002075; NCI-2015-01812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CINJ # 001209; 001209 (Other: Rutgers Cancer Institute of New Jersey); P30CA072720 (NIH); Pro2012002075 (Other: Rutgers)
Record Dates: First submitted 2016-02-17; First posted 2016-02-23 (Estimated); Last update posted 2023-08-07 (Actual); Status verified 2023-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ancillary-Correlative (genomic analysis): Previously collected tissue samples are analyzed for the presence of mutations via next generation sequencing. Patients may also undergo collection of blood samples for analysis of circulating cell-free DNA and circulating tumor cells.
  Interventions: Other: Cytology Specimen Collection Procedure; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Other: Cytology Specimen Collection Procedure — Undergo collection of blood samples
  Other Names: Cytologic Sampling
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This research trial studies the use of targeted genomic analysis of blood and tissue samples from patients with cancer. Genomic sequencing is a laboratory method that is used to determine the entire genetic makeup of a specific organism or cell type. Genomic sequencing can be used to find changes in areas of the genome that may be important in the development of cancer. It may also help doctors improve ways to diagnose and treat patients with rare cancers with poor prognosis or lack of effective therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain blood and tumor tissue for next-generation sequencing and determine the frequency of finding genomic alterations for which there are clinically available (commercially or research based) targeted therapies. Treating clinicians will be provided with relevant validated mutation data for treatment or referral of the patient to pertinent studies.

II. To collect clinical outcomes of patients with actionable mutations for which sequencing has been performed.

III. To obtain tumor genome data for data storage and future computational analysis and correlation with clinical data.

IV. To obtain tumor tissue for development of future in vitro and in vivo cancer models.

OUTLINE:

Previously collected tissue samples are analyzed for the presence of mutations via next generation sequencing. Patients may also undergo collection of blood samples for analysis of circulating cell-free deoxyribonucleic acid (DNA) and circulating tumor cells.

After completion of study, patients are followed up every 3 months for 2 years and then every 6 months for 15 years.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky/Lansky performance score >= 30
* A signed written informed consent
* Evaluation in surgical/medical/radiation oncology/radiology clinic, with a history of biopsy-confirmed diagnosis of cancer of rare histology and/or poor prognosis with standard therapy; priority will be given to rare cancers with poor prognosis and lack of effective standard therapy; study principal investigator (PI) or designee will review and approve each case before enrollment
* Paraffin blocks of the patient's tumor tissue are available and accessible for analysis

Exclusion Criteria:

* Karnofsky/Lansky performance score < 30
* Life expectancy < 3 months

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Sampling Method: Non-Probability Sample
Enrollment: 1100 (Estimated)
Dates: Start 2013-02; Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Frequencies of individual specific mutations and combinations of mutations of related pathway genes | Up to 15 years
  Descriptive analysis will be used to determine frequencies of specific mutations and to determine the pathways that can be targeted most frequently in patients with rare/poor prognosis cancer.
Rate of actionable mutations in rare and/or poor prognosis cancers | Up to 15 years
  The actual rate of mutations found in this study will be determined to estimate the true underlying mutation rate.

CONTACTS AND LOCATIONS:
Overall Officials: Shridar Ganesan, Principal Investigator — Rutgers Cancer Institute of New Jersey
Locations (11):
- United States (11):
  - Ocean Medical Center, Brick, New Jersey
  - Bayshore Community Hospital, Holmdel, New Jersey
  - RWJBarnabas Health - Jersey City Medical Center, Jersey City, Jersey City, New Jersey
  - Southern Ocean County Medical Center, Manahawkin, New Jersey
  - Morristown Medical Center, Morristown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Riverview Medical Center, Red Bank, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No